CLINICAL TRIAL: NCT01729858
Title: Factors Influencing the Survival of Implant-Supported All-Ceramic Prostheses
Brief Title: Survival of Implant-Supported All-Ceramic Prostheses
Status: Active, not recruiting | Type: Observational
Sponsor: University of Florida (Other)
Collaborators: National Institute of Dental and Craniofacial Research (NIDCR) (NIH); Ivoclar Vivadent AG (Industry); Dentsply Sirona Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: IRB201601767-N
Record Dates: First submitted 2012-11-14; First posted 2012-11-20 (Estimated); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Partial Edentulism; Disorder of Prostheses and Implants; Dental Prosthesis Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Device: Yes

GROUPS / COHORTS (2):
- Metal-Ceramic: Metal Ceramic prosthesis with press on veneer with different thicknesses, different diameters of curvature of gingival embrasure and connector heights.
  Interventions: Device: Metal-Ceramic
- Ceramic-Ceramic: Zirconia computer aided design and computer milled cores with press on veneers with different thicknesses, gingival embrasure diameters and connector heights.
  Interventions: Device: Ceramic-Ceramic

INTERVENTIONS:
Device: Ceramic-Ceramic — Zirconia computer aided design and computer milled cores with press on veneers with different thicknesses, gingival embrasure diameters and connector heights.
  Fifty percent of the recruited subjects will be given a ceramic-ceramic bridge at baseline.
  Groups: Ceramic-Ceramic
Device: Metal-Ceramic — Metal Ceramic prosthesis with press on veneer with different thicknesses, different diameters of curvature of gingival embrasure and connector heights.
  Fifty percent of the recruited subjects will receive the metal-ceramic bridges at baseline.
  Groups: Metal-Ceramic

SUMMARY:
The purpose of this research study is to identify reasons that cause an all-ceramic bridge to fracture which include the thickness of the bridge material, the type of bridge material and the bite force of the person. This all-ceramic bridge will be compared to a metal-ceramic bridge. The investigators are conducting this study so we can make bridges which can withstand forces in the mouth which tend to break them.

The overall objective of this research is to analyze how properties of ceramic materials and different forces in the mouth interact with each other to affect the longevity of these bridges. These include fracture toughness, elastic modulus of ceramic layers and supporting substrate, core thickness, connector height, wear, loading orientation, and maximum clenching force.

DETAILED DESCRIPTION:
The long-range goal of the proposed research is to formulate design survival statistics that will aid the dental community in fabricating properly designed prostheses that can predictably survive the oral environment.

Patients who qualify for this study will be randomized (as in chanced with the flip of a coin) into two groups. The first group is a metal-ceramic group where patients will receive a bridge with a metal substructure underneath. The second group is an all-ceramic group where patients will receive a bridge which is made of hard ceramic material. All patients will receive two dental implants which will bond to bone for a period of 4-6 months. An impression or mold of the implants will then be made and a bridge will be fabricated based on the randomization of the patient. Patients will be asked to return at 6 months and yearly thereafter up to 5 years. During these recall appointments, photographs will be taken and impressions of the bridge and other teeth will be made. This will allow us to measure the amount of wear happening with the bridge and the other teeth. The investigators can also examine the amount of bone around the implants as well as the integrity of the bridge.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 21-75 years, and no contraindications to dental treatment.
* Good overall dental health, no active caries, no periodontal disease, and periodontal pocket depths not greater than 4 mm.
* Missing at least three teeth in the posterior area of the mouth.
* Natural teeth opposing the edentulous area and a full complement of teeth or restored teeth in all other areas of the mouth
* Adequate bone height and width at areas of proposed implant sites
* Adequate interocclusal distance to accommodate prosthesis
* Good oral hygiene and compliance with oral hygiene instructions as determined by the amount of plaque present on tooth surfaces.
* Compliance with appointments and willing to pay $2625 for a 3-unit implant supported FDP

Exclusion Criteria:

Non compliance Not enough teeth remaining Uncontrolled medical condition

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients accessing a dental clinic for bridge placement
Sampling Method: Non-Probability Sample
Enrollment: 106 (Actual)
Dates: Start 2008-12 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Fracture | A change from baseline to year 5
  Any fracture or chipping of the prostheses reported by the participant or noted at recall periods

SECONDARY OUTCOMES:
Wear of prosthesis and enamel antagonist | 6 mos, 1 year, 2 year, 3 year, 4 year, 5 year
  Wear of the prosthesis and the opposing enamel will be assessed at the recall appointments

CONTACTS AND LOCATIONS:
Overall Officials: Josephine F Esquivel-Upshaw, DMD,MS,MS-CI, Principal Investigator — University of Florida; Kenneth J Anusavice, PhD, DMD, Study Director — University of Florida; Arthur E Clark, PhD, DMD, Study Director — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

REFERENCES:
- [Background] Esquivel-Upshaw J, Mehler A, Clark A, Neal D, Gonzaga L, Anusavice K. Peri-implant complications for posterior endosteal implants. Clin Oral Implants Res. 2015 Dec;26(12):1390-6. doi: 10.1111/clr.12484. Epub 2014 Sep 27. PMID 25263400
- [Background] Esquivel-Upshaw JF, Mehler A, Clark AE, Neal D, Anusavice KJ. Fracture analysis of randomized implant-supported fixed dental prostheses. J Dent. 2014 Oct;42(10):1335-42. doi: 10.1016/j.jdent.2014.07.001. Epub 2014 Jul 9. PMID 25016139
- [Result] Esquivel-Upshaw JF, Clark AE, Shuster JJ, Anusavice KJ. Randomized clinical trial of implant-supported ceramic-ceramic and metal-ceramic fixed dental prostheses: preliminary results. J Prosthodont. 2014 Feb;23(2):73-82. doi: 10.1111/jopr.12066. Epub 2013 Jun 12. PMID 23758092
- [Derived] Esquivel-Upshaw JF, Mecholsky JJ Jr, Clark AE, Jenkins R, Hsu SM, Neal D, Ren F. Factors influencing the survival of implant-supported ceramic-ceramic prostheses: A randomized, controlled clinical trial. J Dent. 2020;103S:100017. doi: 10.1016/j.jjodo.2020.100017. Epub 2020 Apr 17. PMID 34059304
- [Derived] Mecholsky JJ, Hsu SM, Jadaan O, Griggs J, Neal D, Clark AE, Xia X, Esquivel-Upshaw JF. Forensic and reliability analyses of fixed dental prostheses. J Biomed Mater Res B Appl Biomater. 2021 Sep;109(9):1360-1368. doi: 10.1002/jbm.b.34796. Epub 2021 Feb 1. PMID 33527747